CLINICAL TRIAL: NCT00785707
Title: Littlears Auditory Questionnaire Validation Study in CI Children With LittlEARS My Diary: Language: North American English
Brief Title: Littlears Auditory Questionnaire: Validation Study in CI Children
Acronym: LittlEars
Status: Completed | Type: Observational
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EL NA 020
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Hearing Loss
Keywords: sensorineural hearing loss; cochlear implant
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cochlear implant: children less than 24 months at time of cochlear implantation

SUMMARY:
The LittlEARS Auditory Questionnaire is designed to assess the development of the auditory behavior in children during the first two (hearing) years. The questionnaire has been validated on children with normal hearing whose native language is German. A comparison was made between North American English speaking children with normal hearing and found that it was consistent with the German data. This study is to validate the questionnaire in children with cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

General:

* Less than or 24 months of age prior to implantation
* Cochlear implant candidate deemed by the clinic
* To be implanted with a MED-EL cochlear implant PULSARCI100 or SONATATI100
* English as the primary language at home
* Realistic expectations of guardians
* Willing and available to comply with all scheduled procedures as defined in the protocol

Medical:

* Good general health status, as judged by Primary Investigator
* No contraindications for surgery, in general, or cochlear implant surgery in particular

Exclusion Criteria:

General:

* Prior experience with any cochlear implant system
* Older than 24 months at time of implantation

Medical:

* Severed or non-functional auditory nerve in the ear(s) to be implanted
* Cognitive and/or neurological dysfunction

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 24 months at time of cochlear implantation recommended by the cochlear implant clinic.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2008-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Georgia Health Sciences University, Augusta, Georgia
  - University of North Carolina-Chapel Hill/CCCDP, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Fisseni HJ. (1998) Lehrbuch der psychologischen Diagnostik, Göttingen, Hogrefe.
- [Background] Kühn-Inacker H, Weichbold V, Tsaikpini L, Coninx F, D'Hease P. (2003) LittlEARS Hörfragebogen - Handanweisung. MED-EL Headquarters, Innsbruck, Austria.
- [Background] Weichbold V, Tsiakpini L, Coninx F, D'Haese P. [Development of a parent questionnaire for assessment of auditory behaviour of infants up to two years of age]. Laryngorhinootologie. 2005 May;84(5):328-34. doi: 10.1055/s-2004-826232. German. PMID 15909244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cochlear Implant
Started | 31
Completed | 24
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: months] | 16.2 [11.1 to 24.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: To Validate the LittleEARS Auditory Questionnaire
Description: The LittleEARS auditory questionnaire (LEAQ) uses parent responses to assess auditory behavior in children up to 24 months of age. The questionnaire is scored from 0 to 35 with 0 indicating poorer performance and 35 indicating better performance. There are no subscales for the questionnaire.
Time Frame: 24 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 24
units on a scale | 34.75 [33 to 35]

2. Secondary Outcome: Change in LEAQ Scale Score of Cochlear Implanted Children Over 24 Months After First CI Fitting
Description: The LittleEARS auditory questionnaire (LEAQ) uses parent responses to assess auditory behavior in children up to 24 months of age. The questionnaire is scored from 0 to 35 with 0 indicating poorer performance and 35 indicating better performance. There are no subscales for the questionnaire. This outcome measure is reported as a change on the LEAQ scale from initial CI fitting to 24 months.
Time Frame: 24 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 24
units on a scale | 28.78 [10 to 35]

ADVERSE EVENTS:
Arm/Group | Cochlear Implant
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No